CLINICAL TRIAL: NCT00803777
Title: In-Clinic and Home-Use Study of the AVATAR Blood Glucose Monitoring System in Children and Young Adults
Brief Title: In-Clinic and Home-Use Study of a New Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2008-23
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2010-06-16 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Subjects with type 1 diabetes and healthcare professionals (HCP) used a new blood glucose monitoring system (BGMS) with subject capillary blood. Any subject under age 18 was accompanied by a parent or guardian, who assisted subject if applicable.
  Interventions: Device: Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Investigational Blood Glucose Monitoring System — Subjects with diabetes used a new blood glucose monitoring system with capillary blood. Certain results were compared to a laboratory glucose method.

SUMMARY:
The purpose of this study is to evaluate the performance and acceptability of a new blood glucose meter.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age 4 to 24 years
* Routinely performs blood glucose testing at home, at least 2 times per day, for one month or more before enrollment
* Has used a handheld game system to play video games within a year of enrollment
* If above age 18, subject is able to speak, read, and understand English. If below age 18, subject's parent/guardian is able to speak, read, and understand English, and is able to provide appropriate supervision.
* Is willing to complete all study procedures, with appropriate parent/guardian supervision

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Taking prescription anticoagulants (such as Warfarin or heparin) or has clotting problems that may prolong bleeding. Taking Plavix or aspirin daily is not excluded
* Infection with a blood borne pathogen (e.g., HIV, hepatitis)
* Subject or parent/guardian is employee of competitive medical device company
* Cognitive disorder or other condition, which in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study

Ages: 4 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Aisenberg, MD, Principal Investigator — Hackensack Meridian Health; Georgeanna Klingensmith, MD, Principal Investigator — Barbara Davis Center; Francine Kaufman, MD, Principal Investigator — Children's Hospital Los Angeles; Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Barbara Davis Center, Aurora, Colorado
  - Hackensack University Medical Center, Hackensack, New Jersey

REFERENCES:
- [Result] Parkes JL, Slatin SL, Pardo S, Ginsberg BH. A new consensus error grid to evaluate the clinical significance of inaccuracies in the measurement of blood glucose. Diabetes Care. 2000 Aug;23(8):1143-8. doi: 10.2337/diacare.23.8.1143. PMID 10937512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects actually recruited ranged in age from 5 to 24 years old. Subjects under age 18 were accompanied by a parent or guardian.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 147
Completed | 147
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 147
Age, Customized [Number; unit: participants]
  4-12 years of age | 55
  13-17 years of age | 54
  18-24 years of age | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Duplicate Capillary Results Within +/- 15mg/dL or +/- 20% of Laboratory Glucose Method
Description: Subjects with diabetes (or parents/guardians) and healthcare professionals (HCPs) used a new blood glucose monitoring system (BGMS) with subject capillary blood. BGM results were compared to a lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were obtained in duplicate from subjects(158 BG results possible). The number of capillary results within +/- 15mg/dL (for reference blood glucose values <75mg/dL) or +/- 20% (for reference blood glucose values >/= 75mg/dL)of the reference results were calculated.
Time Frame: 1-2 hours
Population: Some subjects >=13 years old consented to provide larger capillary samples for YSI glucose analysis. Subjects and HCPs provided duplicate results, but one subject's HCP provided only one glucose result. One subject sample was too small to run the YSI analysis; another subject was given carbohydrate to prevent low blood sugar (no results obtained)
Measure: Number; unit: number of capillary results (n=79x2)
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 79
number of capillary results (n=79x2)
  Subjects' Test Results (n=158) | 142
  HCP Test Results (n=157) | 143

2. Primary Outcome: Number of Duplicate Subject BGM Results Within +/- 15mg/dL or +/- 20% of Healthcare Professional Capillary Results
Description: Duplicate subject Blood Glucose Monitoring System (BGMS) results were compared to healthcare professional (HCP) BGMS results (possible number of results = 292). The number of Subject BGM results within +/- 15mg/dL (for reference BG values <75mg/dL) and within +/- 20% (for reference BG values >= 75mg/dL)of the HCP results was calculated.
Time Frame: 1-2 hours
Population: One subject's results were not used because the subject was given carbohydrate to prevent low blood sugar.
Measure: Number; unit: number of Subject BGM Results (n=146x2)
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 146
number of Subject BGM Results (n=146x2) | 277

3. Secondary Outcome: Numbers of BG Results in Zones of the Parkes Error Grid of Clinical Significance of Inaccuracies
Description: The Parkes Error Grid, developed from a survey of 100 clinicians, plots combinations of BG meter measurements against reference method results. Each (x,y) point on the grid is within a risk category, assigned by the clinicians surveyed. Risk categories (increasing severity): ZoneA: No effect on clinical action; ZoneB: Altered clinical action or little/no effect on clinical outcome; ZoneC: Altered clinical action likely to effect clinical outcome; ZoneD: Altered clinical action could have significant medical risk; ZoneE: Altered clinical action could have dangerous consequences
Time Frame: 1-2 hours
Population: Some subjects >=13 yrs consented to provide larger capillary samples for YSI glucose analysis. One subject's sample was insufficient to run the YSI analysis. Another subject's results were not useable as the subject was given carbohydrate to prevent low blood sugar. Duplicate subject BG results provided 158 possible data points.
Measure: Number; unit: Number of BG results in zone (n=79x2)
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 79
Number of BG results in zone (n=79x2)
  Zone A | 146
  Zone B | 11
  Zone C | 1
  Zone D | 0
  Zone E | 0

4. Secondary Outcome: Number of Participants Rated as <=2 (Labeling Comprehension)
Description: Subjects or parents/guardians, as applicable, performed meter tasks after reading the User Guide and Quick Reference Guide. The study staff rated the participants on their success at performing the tasks as follows:
  1. Successful in performing tasks correctly without assistance
  2. Successful after study staff prompted participant to review User Guide.
  3. Successful after study staff assisted subject. (Similar to review of a specific function during a Customer Service call.)
  4. Subject did not perform task correctly and study staff intervention was required.
Time Frame: 1-2 hours
Population: For 2 different subjects, study staff did not rate subject success at 1 task.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 147
participants
  Turn meter on and off (n=147) | 147
  Set time and date (n=147) | 137
  Put strip into the meter (n=146) | 146
  Run control solution (n=146) | 144
  Switch from level 1 to level 2 features (n=147) | 135

5. Secondary Outcome: Average Within Replicate Coefficient of Variation CV (Precision)
Description: The average Coefficient of Variation (CV) was computed by calculating the square of the CV for each pair of Blood Glucose (BG) self-test results, averaging this square value over the number of subjects included in the analysis, and then taking the square root.
Time Frame: 1-2 hours
Population: Meter results were used from subject and HCP data that had numeric values for duplicate BG self-tests. One subject data set was not used because subject was given carbohydrate to prevent low blood sugar. Two subjects' meter results contained outliers (NCCLS EP-9A) and one HCP's results had only one replicate result so these sets were not analyzed.
Measure: Number; unit: percentage CV
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 145
percentage CV
  Average Subject (144) Coefficient of Variation CV | 5.9
  Average HCP (145) Coefficient of Variation CV | 7.2

ADVERSE EVENTS:
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 0/147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less